CLINICAL TRIAL: NCT04386603
Title: Risk Factors for Postoperative Shoulder-tip Pain After Laparoscopic Surgery Undergoing General Anesthesia
Status: Completed | Type: Observational
Sponsor: Shenzhen Second People's Hospital (Other)
Collaborators: Shenzhen Third People's Hospital (Other)
Responsible Party: Principal Investigator, ZhiHeng Liu, Head of Anesthesiology, Shenzhen Second People's Hospital
Other Study IDs: KS20190903004-FS02
Record Dates: First submitted 2020-05-04; First posted 2020-05-13 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Laparoscopic Surgery; Anesthesia
Keywords: risk factor; laparoscopic surgery; postoperative shoulder pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- shoulder-tip pain group: The patients in this group have postoperative phoulder-tip pain after laparoscopic surgery undergoing general anesthesia.
- non-shoulder-tip pain group: The patients in this group don't have postoperative phoulder-tip pain after laparoscopic surgery undergoing general anesthesia.

SUMMARY:
To find out the risk factors for postoperative shoulder-tip pain after laparoscopic surgery undergoing general anesthesia.

DETAILED DESCRIPTION:
To find out the risk factors for postoperative shoulder-tip pain after laparoscopic surgery undergoing general anesthesia.Besides,this research also aims to observe the incidence of postoperative shoulder-tip pain after laparoscopic surgery undergoing general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years old (including 18 years old) having gynecologic or gastrointestinal or hepatobiliary surgery undergoing general anesthesia;
2. Patients agreeing to participate in the study and sign the informed consent.

Exclusion Criteria:

1. Patients under 18 years age or having emergency laparoscopic surgery;
2. Patients having laparoscopy but not undergoing general anesthesia;
3. Patients undergoing laparoscopy and having hysteroscopy at the same time.
4. Patients undergoing laparoscopy and having fistulostomy at the same time.
5. Patients having regional thermoperfusion after laparoscopic surgery.
6. Laparoscopy being needed to converse to laparotomy.
7. Patients having shoulder pain or history of periarthritis of shoulder or long-term taking painkillers.
8. Patients having severe psychological problem and unable to cooperate with our study.
9. Patients being sent to ICU for further treatment after operation.
10. Patients being discharged within 2 days after operation and losing contact.
11. Patients having another operation after laparoscopy.
12. Patients taking another painkillers except using patient-controlled intravenous analgesia.
13. Patients refusing to take part in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included in this research all have diseases which need to have surgeries to fix their problems.Some of them not only have one disease but have two or more diseases such as cardiovascular disfunction,respiratory disfunction and so on.All of them are Asian and over 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 1311 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
inpatient department | Baseline (before laparoscopic surgery)
  Compare the inpatient department difference between two groups.The inpatient department include the department of gynecology, gastrointestinal surgery and hepatolugical surgery.The investigators read the medical record to find out which department the patient is in.
sex | Baseline (before laparoscopic surgery)
  Compare sex(male or female)difference between two groups.
age | Baseline (before laparoscopic surgery)
  Compare age difference between two groups.
body mass index(BMI) | Baseline (before laparoscopic surgery)
  Compare BMI difference between two groups.First,investigators get the weight(kg）and height(m) of the patient from medical record.Then BMI(kg/m^2) is calculated with the formula,weight(kg)/height(m)^2.
ASA grade | Baseline (within laparoscopic surgery)
  Compare ASA grade difference between two groups.The ASA grade includes five grades(Ⅰ,Ⅱ,Ⅲ,Ⅳ,Ⅴ）.The investigators collect this information from the anesthesia record.
operative position | within laparoscopic surgery
  Compare operative position difference between two groups.The operative position include lateral position,trendelenburg position and feet-down tilt position.The investigators collect this information from the anesthesia record.
peritoneal drainage | within laparoscopic surgery
  Compare the use of peritoneal drainage difference(used or unused) between two groups.The investigators collect this information from operation record.
operative duration | within laparoscopic surgery
  Compare operative duration(minutes) between two groups.The investigators collect this information from operation record.
the use of sufentanil | within laparoscopic surgery
  Compare the use of sufentanil difference(used or unused)between two groups.The investigators collect this information from the anesthesia record.
the use of fentanyl | within laparoscopic surgery
  Compare the use of fentanyl difference(used or unused) between two groups.The investigators collect this information from the anesthesia record.
the use of remifentanil | within laparoscopic surgery
  Compare the use of remifentanil difference(used or unused) between two groups.The investigators collect this information from the anesthesia record.
the use of morphine | within laparoscopic surgery
  Compare the use of morphine difference(used or unused) between two groups.The investigators collect this information from the anesthesia record.
the use of butophanol | within laparoscopic surgery
  Compare the use of butophanol difference(used or unused) between two groups.The investigators collect this information from the anesthesia record.
the use of sevoflurane | within laparoscopic surgery
  Compare the use of sevoflurane difference(used or unused) between two groups.The investigators collect this information from the anesthesia record.
the use of flubiprofen | within laparoscopic surgery
  Compare the use of flubiprofen difference(used or unused) between two groups.The investigators collect this information from the anesthesia record.
the use of parecoxib | within laparoscopic surgery
  Compare the use of parecoxib difference(used or unused) between two groups.The investigators collect this information from the anesthesia record.
the use of dezocine | within laparoscopic surgery
  Compare the use of dezocine difference(used or unused) between two groups.The investigators collect this information from the anesthesia record.
the use of tramadol | within laparoscopic surgery
  Compare the use of tramadol difference(used or unused) between two groups.The investigators collect this information from the anesthesia record.
the use of intravenous lidocaine | within laparoscopic surgery
  Compare the use of intravenous lidocaine difference(used or unused) between two groups.The investigators collect this information from the anesthesia record.
the use of dexamethasone | within laparoscopic surgery
  Compare the use of dexamethasone difference(used or unused) between two groups.The investigators collect this information from the anesthesia record.
the use of methylprednisolone | within laparoscopic surgery
  Compare the use of methylprednisolone difference(used or unused) between two groups.The investigators collect this information from the anesthesia record.
the use of deep neuromuscular block | within laparoscopic surgery
  Compare the use of deep neuromuscular block difference(used or unused) when undergoing general anesthesia between two groups.Neuromuscular block was monitored using post-tetanic-count(PTC) stimulation by a muscle relaxation monitor.If the PTC is within 1-2,the neuromuscular block of patient is deep.If not, the neuromuscular block of patient is not deep.The investigators collect this information from the anesthesia record.
the use of peripheral nerve block | within laparoscopic surgery
  Compare the use of peripheral nerve block difference(used or unused) when undergoing general anesthesia between two groups.The types of peripheral nerve block in our study include ilioinguinal and iliohypogastric nerve blocks,transversus abdominis plane block(TAP) and rectus sheath block(RSB).Patients who using any kind of the above peripheral nerve block belong to the group that is using peripheral nerve block when undergoing general anesthesia.The investigators collect this information from the anesthesia record.
the use of tracer-site infiltration with ropinvacaine | within laparoscopic surgery
  Compare the use of tracer-site infiltration with ropinvacaine difference(used or unused) when undergoing general anesthesia between two groups.The investigators collect this information from the anesthesia record.
the use of patient-controlled intravenous analgesia | two days after laparoscopic surgery
  Compare the use of patient-controlled intravenous analgesia(PCIA) difference(used or unused) after laparoscopic surgery.The drugs for patients using PCIA to control pain are different but the investigators ignore the difference of the drug composition.As long as the patient uses PCIA,he or she belongs to the using group.The investigators collect this information from the anesthesia record.

SECONDARY OUTCOMES:
incidence of postoperative shoulder-tip pain after laparoscopic surgery undergoing general anesthesia | two months after laparoscopic surgery
  Calculate and find out the incidence of postoperative shoulder-tip pain after laparoscopic surgery undergoing general anesthesia.First,the investigators pay the follow-up visit to the patients two days after laparoscopy asking them vocally if they have postoperative shoulder-tip pain.Then the investigators count the number of people who have postoperative shoulder-tip pain after laparoscopic surgery(N1) and the number of people who don't have postoperative shoulder-tip pain after laparoscopic surgery(N2).Finally, the incidence of postoperative shoulder-tip pain after laparoscopic surgery undergoing general anesthesia (%)is calculated with the formula,N1/(N1+N2).(N1+N2)is equal to the total number of the patients entering our study.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Zhiheng, Doctor, Study Chair — Anesthesia department of ShenZhen Second People's Hospital
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Song T, Kim KH, Lee KW. The Intensity of Postlaparoscopic Shoulder Pain Is Positively Correlated with the Amount of Residual Pneumoperitoneum. J Minim Invasive Gynecol. 2017 Sep-Oct;24(6):984-989.e1. doi: 10.1016/j.jmig.2017.06.002. Epub 2017 Jun 7. PMID 28602786
- [Result] Jackson SA, Laurence AS, Hill JC. Does post-laparoscopy pain relate to residual carbon dioxide? Anaesthesia. 1996 May;51(5):485-7. doi: 10.1111/j.1365-2044.1996.tb07798.x. PMID 8694166
- [Result] Bogani G, Uccella S, Cromi A, Serati M, Casarin J, Pinelli C, Ghezzi F. Low vs standard pneumoperitoneum pressure during laparoscopic hysterectomy: prospective randomized trial. J Minim Invasive Gynecol. 2014 May-Jun;21(3):466-71. doi: 10.1016/j.jmig.2013.12.091. Epub 2013 Dec 25. PMID 24374246
- [Result] Hsu KF, Chen CJ, Yu JC, Wu SY, Chen BC, Yang CW, Chen TW, Hsieh CB, Chan DC. A Novel Strategy of Laparoscopic Insufflation Rate Improving Shoulder Pain: Prospective Randomized Study. J Gastrointest Surg. 2019 Oct;23(10):2049-2053. doi: 10.1007/s11605-018-3896-5. Epub 2018 Oct 8. PMID 30298416
- [Result] Williams WH 3rd, Cata JP, Lasala JD, Navai N, Feng L, Gottumukkala V. Effect of reversal of deep neuromuscular block with sugammadex or moderate block by neostigmine on shoulder pain in elderly patients undergoing robotic prostatectomy. Br J Anaesth. 2020 Feb;124(2):164-172. doi: 10.1016/j.bja.2019.09.043. Epub 2019 Nov 26. PMID 31780139
- [Result] Wada S, Fukushi Y, Nishimura M, Matsumoto S, Takimoto K, Imai K, Ota H, Tsuzuki Y, Nakajima A, Fujino T. Analysis of risk factors of postlaparoscopic shoulder pain. J Obstet Gynaecol Res. 2020 Feb;46(2):310-313. doi: 10.1111/jog.14156. Epub 2020 Jan 20. PMID 31958892
- [Result] Donatsky AM, Bjerrum F, Gogenur I. Surgical techniques to minimize shoulder pain after laparoscopic cholecystectomy. A systematic review. Surg Endosc. 2013 Jul;27(7):2275-82. doi: 10.1007/s00464-012-2759-5. Epub 2013 Jan 24. PMID 23340814